CLINICAL TRIAL: NCT05896670
Title: A Multi-center, Randomized, Double-Masked, Vehicle-Controlled Study Evaluating the Efficacy and Safety of Licaminlimab for the Treatment of Dry Eye Disease
Brief Title: Safety and Efficacy of Licaminlimab Ophthalmic Solution for the Treatment of Dry Eye Disease
Acronym: RELIEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oculis (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC-201
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Disease
Keywords: Ophthalmology; Topical Ophthalmic Solution; Eye Drop; DED
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- licaminlimab (OCS-02) (Experimental): 60 mg/mL licaminlimab ophthalmic solution
  Interventions: Drug: licaminlimab; Other: Artificial tears
- Vehicle (Placebo Comparator): Vehicle of licaminlimab (OCS-02) ophthalmic solution
  Interventions: Other: vehicle of OCS-02; Other: Artificial tears

INTERVENTIONS:
Drug: licaminlimab — ophthalmic solution 60 mg/mL Subjects will be randomized to receive licaminlimab eye drops three times daily (TID) for 6 weeks.
  Other Names: OCS-02
  Arms: licaminlimab (OCS-02)
Other: vehicle of OCS-02 — inert ophthalmic solution vehicle of OCS-02 Subjects will be randomized to receive vehicle eye drops three times daily (TID) for 6 weeks.
  Arms: Vehicle
Other: Artificial tears — Subjects who quality after an initial screening were entered into a run-in phase where they received artificial tears to use three times daily (TID) for approximately 14 days.

SUMMARY:
The goal of this clinical trial is to learn about licaminlimab (OCS-02) in the treatment of dry eye disease. The main question it aims to answer is if licaminlimab ophthalmic solution is more effective than vehicle in treating signs of dry eye disease.

DETAILED DESCRIPTION:
This is a Phase 2b, multicenter, randomized, double-masked, vehicle-control study designed to evaluate the efficacy and safety of licaminlimab for the treatment of signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Provide written informed consent.
* Be willing and able to comply with all study procedures.
* Have a history of dry eye disease for at least 6 months prior to Visit 1.

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at least one eye at Visit 1 that may include active blepharitis, meibomian gland dysfunction, lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the Investigator may interfere with study parameters.
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation in at least one eye at Visit 1 or Visit 2.
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses in the study eye during the study.

  * Additional inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of licaminlimab in subjects with signs of dry eye disease | Baseline to Day 43
  Endpoints of signs of dry eye disease (staining, redness, Schirmer's test) at various time points throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Klier, MD, MPH, Study Director — Oculis
Locations (5):
- United States (5):
  - Oculis Investigative Site, Newport Beach, California
  - Oculis Investigative Site, Colorado Springs, Colorado
  - Oculis Investigative Site, Shelby, North Carolina
  - Oculis Investigative Site, Erie, Pennsylvania
  - Oculis Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No